CLINICAL TRIAL: NCT02651415
Title: A Phase II Trial of the Effect of Perindopril on HFSR Incidence and Severity in Patients Receiving Regorafenib With Refractory Metastatic Colorectal Carcinoma (mCRC)
Brief Title: Phase II Study of Perindopril and Regorafenib in mCRC
Acronym: PARICCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H15-02424
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Metastatic colorectal carcinoma; mCRC; Regorafenib; Stivarga; Perindopril; Perindopril erbumine; Coversyl
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib and Perindopril (Experimental): Phase II, open label, single arm trial of patient with refractory mCRC treated with regorafenib (10 mg/day) and perindopril (4 mg/day). There will be no stratification in this study.
  Interventions: Drug: Regorafenib; Drug: Perindopril

INTERVENTIONS:
Drug: Regorafenib — Stivarga® will be used as per the marketed indication ("on label"), Coversyl will be used off-label and as such a Clinical Trial Application will be filed with Health Canada.
  Regorafenib will be administered 160 mg daily for 21 days of a 28 day cycle. Regorafenib will be administered with low fat breakfast, one hour after perindopril. A low fat breakfast as defined by the Stivarga ® (regorafenib) Product Monograph is one that is <30% fat, ~300-550 calories.
  Other Names: Stivarga (regorafenib) or "regorafenib"
Drug: Perindopril — COVERSYL® (perindopril erbumine) 4 mg will be administered daily for 21 days of a 28 day cycle. Perindopril will be administered orally, first thing in the morning on an empty stomach.
  Other Names: COVERSYL (perindopril erbumine) or "perindopril"

SUMMARY:
The purpose of this study is to find out what effects the combination of regorafenib and perindopril has on hand-foot skin reaction (HFSR), on high blood pressure (hypertension) and on any other types of side-effects and compare it to the published incidence of the side-effects with regorafenib alone.

This research is being done in an attempt to reduce the side-effects associated with regorafenib.

DETAILED DESCRIPTION:
The investigators hypothesize that treatment of regorafenib-treated mCRC patients with perindopril may reduce HFSR compared to reported incidence and severity.

The investigators also hypothesize that treatment of regorafenib-treated mCRC patients with perindopril will likely reduce hypertension, a known adverse effect of vascular endothelial growth factor/receptor (VEGF/VEGFR) inhibition.

According to the 2014 Canadian Cancer Statistics, colorectal cancer is the second most frequently diagnosed cancer in Canadian males and the third most frequently diagnosed cancer in Canadian females, accounting for 13.9% and 11.6% of new diagnoses, respectively. Although mortality rates are declining very slightly, colorectal cancer is the second most frequent cause of cancer deaths in males and the third most frequent cause of cancer death in females, at 12.8% and 11.5% respectively.

Metastatic colorectal cancers are generally not curable. Median overall survival for patients with unresectable mCRC who receive best supportive care (BSC) is five to six months. Palliative treatment with systemic chemotherapy is the best option prolonging survival and maintaining quality of life. Patients who are exposed to all active drugs can sometimes extend survival past two years.

For many years 5 Fluorouracil (FU) was the only treatment, but the approval of irinotecan, oxaliplatin, fluoropyrimidines, as well as various monoclonal antibodies targeting VEGF and epidermal growth factor receptor (EGFR) growth factors led to the development of a number of different regimens. The ideal combination and sequence of the different agents is still not determined.

Recently, Regorafenib has shown efficacy in patients pretreated with all these options in a large phase III trial, where it prolonged overall survival (OS) compared with placebo (Grothey, et al 2013). In addition, the results were confirmed in a smaller randomised trial in the Asian population, with patients being less intensively pre-treated (Li et al, 2014). Therefore, regorafenib is now considered a standard option in pre-treated patients.

The intended outcome of successfully and significantly mitigating regorafenib-induced HFSR is that patients will be able to stay on the regorafenib for a longer period to increase efficacy. The hypothesis underlying this trial is that the co-administration of perindopril with regorafenib will mitigate HFSR symptoms.

This may not be the case, and if the HFSR is more severe with the addition of perindopril than with regorafenib alone, the study will be discontinued.

As a secondary endpoint, hypertension will also be followed.

ELIGIBILITY:
Inclusion Criteria:

Patients with metastatic colorectal cancer (mCRC) who have progressed on/after, or are intolerant to all approved drugs for CRC and are eligible for regorafenib.

In order to be eligible, all inclusion criteria must be met.

A patient must:

* Understand, be willing to give consent, and sign a written informed consent form (ICF) prior to undergoing any study-specific procedure
* Be male or female and ≥ 18 years of age
* Histological or cytological documentation of adenocarcinoma of the colon or rectum.
* Patients with metastatic colorectal cancer (Stage IV) previously treated with fluoropyrimidine-based chemotherapy, oxaliplatin, irinotecan, an anti-VEGF therapy, and, if KRAS wild type, an anti-EGFR therapy.
* Progression during or within 3 months following the last administration of approved standard therapies, or have experienced intolerance to previous therapy.
* Metastatic CRC patients with measurable or non-measurable disease
* Life expectancy of at least 3 months
* Have an Eastern Cooperative Oncology Group performance status of 0 or 1 (within 14 days prior to the initiation of study treatment)
* Have adequate bone marrow, liver function, and renal function as measured by the following laboratory assessments conducted within 7 days prior to the initiation of study treatment:

  * Total bilirubin < 1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 times the ULN (< 5 times ULN for patients with liver involvement of their cancer)
  * Lipase < 1.5 times the ULN
  * Serum creatinine < 1.5 times the ULN
  * Glomerular filtration rate > 30 mL/min/1.73 m2 according to the modified diet in renal disease abbreviated formula
  * International normalized ratio (INR) of prothrombin time (PT; PT-INR) and partial thromboplastin time (PTT) < 1.5 times the ULN
  * Platelet count > 100000 /mm3, hemoglobin > 9 g/dL, absolute neutrophil count > 1500/mm3.
  * Alkaline phosphatase limit ≤ 2.5 times the ULN (< 5 times ULN for patients with liver involvement of their cancer)
* If female and of childbearing potential, have a NEGATIVE result on a pregnancy test performed a maximum of 7 days before initiation of study treatment.
* If female and of childbearing potential or if male, must agree to use adequate contraception (e.g., abstinence, intrauterine device, oral contraceptive, or double-barrier method) based on the judgment of the investigator or a designated associate from the date on which the ICF is signed until 6 months after the last dose of study drug.

Exclusion Criteria:

Patients who meet the following criteria at the time of screening will be excluded:

* Patients with hypotension (less than 90/60mm Hg) or at risk of symptomatic hypotension (fainting or dizziness) will be excluded.
* Prior treatment with regorafenib or any VEGFR-targeting kinase inhibitor.
* Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.
* Concurrent cancer requiring treatment that is distinct in primary site or histology from colorectal cancer.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Unstable/uncontrolled cardiac disease including: congestive heart failure > New York Heart Association (NYHA) class 2; unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months); myocardial infarction less than 6 months before start of study drug; cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension. (Systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Patients with phaeochromocytoma.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication.
* Ongoing infection > grade 2 NCI-CTCAE version 4.03
* Known history of human immunodeficiency virus (HIV) infection.
* Known history of chronic hepatitis B or C.
* Patients with seizure disorder requiring medication.
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
* History of organ allograft
* Patients with evidence or history of bleeding diasthesis, including patients who have had a transfusion and/or radiographic endoscopic or elective operative interaction to control the bleeding or hemorrhage event within four weeks prior to the study
* Non-healing wound, ulcer, or bone fracture.
* Renal impairment or failure requiring hemo-or peritoneal dialysis.
* Patients with severe hepatic impairment.
* Dehydration NCI-CTC version 4.03 grade > 1.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any illness or medical conditions that are unstable or could jeopardize the safety of the study
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Persistent proteinuria of Common Terminology Criteria (CTC) Grade 3 or higher. Quantification of proteinuria done by urinary protein/creatinine ratio on a random urine sample preferably taken at mid-morning. If protein/creatinine ratio is greater than 30g/mol Creat, then a 24-hour urine protein test should be performed to confirmed Grade 3 or higher proteinuria (> 3.5 g/24 hours).
* Patients unable to swallow oral medications
* Any malabsorption condition
* Unresolved toxicity higher than NCI-CTCAE (version 4.03) Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity ≤Grade 2
* Patients who are hypersensitive to perindopril, as well as those hypersensitive to regorafenib, sorafenib, drugs in the same class or any ingredient in the formulation.
* Patients who cannot tolerate the full dose of perindopril (4 mg) for any reason.
* Patients receiving systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, hormonal therapy and experimental or approved therapies during this trial or within 14 days before starting to receive study medication.

In addition, patients will be excluded for the following reasons (From perindopril monograph).

* Patients with a history of hereditary/idiopathic angioedema, or angioedema related to previous treatment with an angiotensin converting enzyme inhibitor.
* Pregnant women or those planning to become pregnant, nursing women.
* Patients with hereditary problems of galactose intolerance, glucose-galactose malabsorption, or the Lapp lactase deficiency.
* Patients with pre-existing anti-hypertension treatment with an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) are to be excluded. Co-administration of ACE inhibitors, including COVERSYL®, with other agents blocking the Renin-Angiotensin System (RAS), such as ARBs or aliskiren-containing drugs, will not be allowed, since such treatment has been associated with an increased incidence of severe hypotension, renal failure, and hyperkalemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Renouf, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Anderson TJ, Elstein E, Haber H, Charbonneau F. Comparative study of ACE-inhibition, angiotensin II antagonism, and calcium channel blockade on flow-mediated vasodilation in patients with coronary disease (BANFF study). J Am Coll Cardiol. 2000 Jan;35(1):60-6. doi: 10.1016/s0735-1097(99)00537-9. PMID 10636260
- [Background] Ceconi C, Fox KM, Remme WJ, Simoons ML, Bertrand M, Parrinello G, Kluft C, Blann A, Cokkinos D, Ferrari R; EUROPA Investigators; PERTINENT Investigators and the Statistical Committee. ACE inhibition with perindopril and endothelial function. Results of a substudy of the EUROPA study: PERTINENT. Cardiovasc Res. 2007 Jan 1;73(1):237-46. doi: 10.1016/j.cardiores.2006.10.021. Epub 2006 Nov 10. PMID 17140552
- [Background] Ceconi C, Francolini G, Olivares A, Comini L, Bachetti T, Ferrari R. Angiotensin-converting enzyme (ACE) inhibitors have different selectivity for bradykinin binding sites of human somatic ACE. Eur J Pharmacol. 2007 Dec 22;577(1-3):1-6. doi: 10.1016/j.ejphar.2007.07.061. Epub 2007 Aug 3. PMID 17716647
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Erber R, Thurnher A, Katsen AD, Groth G, Kerger H, Hammes HP, Menger MD, Ullrich A, Vajkoczy P. Combined inhibition of VEGF and PDGF signaling enforces tumor vessel regression by interfering with pericyte-mediated endothelial cell survival mechanisms. FASEB J. 2004 Feb;18(2):338-40. doi: 10.1096/fj.03-0271fje. Epub 2003 Dec 4. PMID 14657001
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Grothey A, George S, van Cutsem E, Blay JY, Sobrero A, Demetri GD. Optimizing treatment outcomes with regorafenib: personalized dosing and other strategies to support patient care. Oncologist. 2014 Jun;19(6):669-80. doi: 10.1634/theoncologist.2013-0059. Epub 2014 May 12. PMID 24821824
- [Background] Li J, Qin S, Yau T et al. CONCUR: a randomized double-blind placebo controlled phase 3 study of regorafenib monotherapy in Asian patients with previously treated metastatic colorectal cancer (mCRC). Ann Oncol 2014; 25 (Suppl 2): ii114-ii115.
- [Background] Miller KK, Gorcey L, McLellan BN. Chemotherapy-induced hand-foot syndrome and nail changes: a review of clinical presentation, etiology, pathogenesis, and management. J Am Acad Dermatol. 2014 Oct;71(4):787-94. doi: 10.1016/j.jaad.2014.03.019. Epub 2014 May 1. PMID 24795111
- [Background] Robert C, Soria JC, Spatz A, Le Cesne A, Malka D, Pautier P, Wechsler J, Lhomme C, Escudier B, Boige V, Armand JP, Le Chevalier T. Cutaneous side-effects of kinase inhibitors and blocking antibodies. Lancet Oncol. 2005 Jul;6(7):491-500. doi: 10.1016/S1470-2045(05)70243-6. PMID 15992698
- [Background] Taddei S: New evidence for entothelial protection. Medicographia, a Servier publication Vol 34:17-23, 2012
- [Background] Zhuo JL, Mendelsohn FA, Ohishi M. Perindopril alters vascular angiotensin-converting enzyme, AT(1) receptor, and nitric oxide synthase expression in patients with coronary heart disease. Hypertension. 2002 Feb;39(2 Pt 2):634-8. doi: 10.1161/hy0202.103417. PMID 11882622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted from August 2016 - November 2018. 12 Patients were enrolled but only 10 were evaluable.
Groups:
- Single Arm Trial: All patients in this single-arm trial will receive treatment with regorafenib and perindopril.
Period: Overall Study
Arm/Group | Single Arm Trial
Started | 12 (12 patients were enrolled.)
Completed | 10 (10 patients were evaluable.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Regorafenib and Perindopril: Phase II, open label, single arm trial of patient with refractory metastatic colorectal carcinoma (mCRC) treated with regorafenib (10 mg/day) and perindopril (4 mg/day). There will be no stratification in this study.
  Regorafenib: Stivarga® will be used as per the marketed indication ("on label"), Coversyl will be used off-label and as such a Clinical Trial Application will be filed with Health Canada.
  Regorafenib will be administered 160 mg daily for 21 days of a 28 day cycle. Regorafenib will be administered with low fat breakfast, one hour after perindopril. A low fat breakfast as defined by the Stivarga ® (regorafenib) Product Monograph is one that is <30% fat, ~300-550 calories.
  Perindopril: COVERSYL® (perindopril erbumine) 4 mg will be administered daily for 21 days of a 28 day cycle. Perindopril will be administered orally, first thing in the morning on an empty stomach.
Arm/Group | Regorafenib and Perindopril
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Number of participants aged less than or equal to 18 years, between 18 and 65 years, and greater than or equal to 65 years. Population: 12 participants were enrolled but only 10 participants were evaluable.
  Participants
    number analyzed (Participants) | 10
    <=18 years | 0
    Between 18 and 65 years | 6
    >=65 years | 4
Age, Continuous [Median (Full Range); unit: Years] — Median age of participants Population: 12 participants were enrolled but only 10 participants were evaluable.
  Years
    number analyzed (Participants) | 10
    (all) | 60.65 [49 to 72]
Sex: Female, Male [Count of Participants; unit: Participants] — Number of male and female participants. Population: 12 participants were enrolled but only 10 participants were evaluable.
  Participants
    number analyzed (Participants) | 10
    Female | 5
    Male | 5
Race/Ethnicity, Customized [Number; unit: participants] — Number of Asian, Black, and Caucasian participants. Population: 12 participants were enrolled but only 10 participants were evaluable.
  participants
    Asian: number analyzed (Participants) | 10
    Asian | 5
    Black: number analyzed (Participants) | 10
    Black | 1
    Caucasian: number analyzed (Participants) | 10
    Caucasian | 4
Region of Enrollment [Number; unit: participants] — Number of participants for which regional information was collected. Population: 12 participants were enrolled but only 10 participants were evaluable.
  participants
    Canada: number analyzed (Participants) | 10
    Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Have Any Grade HFSR Toxicity
Description: The trial will measure the toxicities of HFSR in participants receiving both perindopril and regorafenib using the CTCAE v4.03 criteria.
  The toxicity of HFSR will be expressed based on the number of participants in the study (N=10) who are experiencing HFSR of all grades.
Time Frame: Up to Safety Follow-Up Visit (30 days +/- 7 days after permanently stopping study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: The Number of Participants That Experienced Any Grade of Hypertension as Assessed by CTCAE v4.03 Criteria When Treated With a Combination of Regorafenib and Perindopril
Description: All grades of hypertension will be evaluated using CTCAE v4.03, weekly for the first six weeks while they are on the study drug, then every second week and during the 30-day follow-up period (Post therapy).
Time Frame: Weekly for the first six weeks while on the study drug, then every second week and during the 30-day follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 10
Participants | 6

3. Secondary Outcome: The Number of Participants That Experienced All Grade Toxicities as Assessed by CTCAE v4.03 Criteria When Treated With a Combination of Regorafenib and Perindopril
Description: All grades of adverse events (including HFSR) will be evaluated using CTCAE v4.03, at baseline and at D1 of each cycle while they are on the study drug and during the 30-day follow-up period (Post therapy).
Time Frame: At baseline and at D1 of each cycle while on the study drug and during the 30-day follow-up period
Measure: Number; unit: participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 10
participants | 10

4. Secondary Outcome: Number of Participants With Maximal Severity of HFSR as Assessed by CTCAE v4.03 Criteria When Treated With a Combination of Regorafenib and Perindopril
Description: The number of participants that experienced an HFSR of grade 3 or above as assessed by CTCAE v4.03 criteria when treated with a combination of regorafenib and perindopril.
Time Frame: Up to Safety Follow-Up Visit (30 days +/- 7 days after permanently stopping study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 10
Participants | 5

5. Secondary Outcome: Median Time Course to Development of Worst Grade (Grade 3) HFSR as Assessed by CTCAE v4.03 Criteria When Treated With a Combination of Regorafenib and Perindopril
Description: Median time course for participants to develop worst grade 3 HFSR toxicity is defined as the time (days) from start date of study drug to date of first documented grade 3 HFSR toxicity and will be calculated only for patients who had a HFSR toxicity grade 3.
Time Frame: p to Safety Follow-Up Visit (30 days +/- 7 days after permanently stopping study treatment)
Measure: Median (Full Range); unit: days
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 10
days | 12 [9 to 83]

6. Secondary Outcome: Median Time to Progression Free Survival (PFS)
Description: Median time (in months) to PFS. PFS is defined as the time from start date of study drugs to the date of first documented disease progression (radiological or clinical) or death due to any cause, if death occurs before progression is documented. PFS will be evaluated based on RECIST v1.1 criteria, 20% progression or any new lesion.
Time Frame: From start date of study drugs to the date of first documented disease progression or death due to any cause.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 10
Months | 2.60 [1.74 to 3.61]

ADVERSE EVENTS:
Time Frame: The PARICCA study was conducted from August 2016 to November 2018 and during this time period, adverse event (AE) data were collected. All grades of AE (including HFSR) were evaluated using CTCAE v4.03, at baseline and at D1 of each cycle while they are on the study drug and during the 30-day follow up period (Post therapy).
Arm/Group | Single Arm Trial
All-Cause Mortality (participants affected / at risk) | 10/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=10)
RUQ Abdominal Pain; Pneumonia (Gastrointestinal disorders) | 1 — Right Upper Quadrant (RUQ) Abdominal Pain; Pneumonia
Malignant Neoplasm, Grade 5 (Gastrointestinal disorders) | 1 — Malignant Neoplasm, Grade 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=10)
Hypertension (Vascular disorders) | 6 — Hypertension
Increased AST (Investigations) | 3 — Increased aspartate aminotransferase (AST)
Fatigue (General disorders) | 7 — Fatigue
Abdominal pain (Gastrointestinal disorders) | 5 — Pain, abdomen
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 — Hand-foot skin reaction
Anorexia (Metabolism and nutrition disorders) | 6 — Anorexia
Mucositis oral (Gastrointestinal disorders) | 6 — Oral mucositis (dry mouth, sore throat, mucosal infection)
Diarrhea (Gastrointestinal disorders) | 5 — Diarrhoea
Myalgia (Musculoskeletal and connective tissue disorders) | 5 — Muscle pain (myalgia)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 — Rash or desquamation
Nausea (Gastrointestinal disorders) | 4 — Nausea
Constipation (Gastrointestinal disorders) | 4 — Constipation
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 — Voice changes/hoarse voice
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 — Arthralgia (joint pain)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 — Pain extremity/neuralgia
Urinary tract infection (Infections and infestations) | 3 — Infection (UTI)
Fever (General disorders) | 3 — Fever (pyrexia)
Dry skin (Skin and subcutaneous tissue disorders) | 3 — Dry skin
Vomiting (Gastrointestinal disorders) | 3 — Vomiting
Ascites (Gastrointestinal disorders) | 3 — Ascites
Headache (Nervous system disorders) | 3 — Headache
Pelvic pain (Reproductive system and breast disorders) | 2 — Thigh, groin, pelvic pain
Non-cardiac chest pain (General disorders) | 2 — Non-cardiac chest pain
Back pain (Musculoskeletal and connective tissue disorders) | 2 — Back pain
Rectal pain (Gastrointestinal disorders) | 2 — Rectal/anal pain
Dysphagia (Gastrointestinal disorders) | 2 — Dysphagia (difficulty swallowing)
Localized edema (General disorders) | 2 — Oedema (ankle)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — Dyspnoea (shortness of breath)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 — Dry cough
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 — Erythaema face
Insomnia (Psychiatric disorders) | 1 — Insomnia
Pruritus (Skin and subcutaneous tissue disorders) | 1 — Pruritis (itchy)
Pain (General disorders) | 1 — Pain, soles of feet, toe
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 — Weakness
Chills (General disorders) | 1 — Chills
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 — Nose bleed (epistaxis)
Weight loss (Investigations) | 1 — Weight loss
Paresthesia (Nervous system disorders) | 1 — Paraesthesia
Hypokalemia (Metabolism and nutrition disorders) | 2 — Hypokalaemia
Blood bilirubin increased (Investigations) | 2 — Hyperbilirubinaemia
Alkaline phosphatase increased (Investigations) | 1 — Increased alkaline phosphatase
Lipase increased (Investigations) | 1 — Increased lipase
INR increased (Investigations) | 1 — Elevated international normalized ratio (INR)
Hematuria (Renal and urinary disorders) | 1 — Haematuria
Cramps (leg) (Musculoskeletal and connective tissue disorders) | 1 — Cramps (leg)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 — Haemoptysis (spitting blood)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02651415/Prot_SAP_000.pdf